CLINICAL TRIAL: NCT06266065
Title: Impact of Coronary Sinus Flow Reducer on Coronary Microcirculation and Myocardial Ischemia in Patients With Refractory Angina Pectoris
Brief Title: Impact of Coronary Sinus Flow Reducer on Coronary Microcirculation and Myocardial Ischemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Josko Bulum, MD, PhD, MD, PhD, Principal Investigator, Clinical Hospital Centre Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8.1-23/260-2;02/013AG
Record Dates: First submitted 2024-02-03; First posted 2024-02-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Coronary Sinus Reducer; Myocardial Ischemia; Coronary Microcirculation
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: Single-Center Prospective Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary Sinus Reducer (Experimental)
  Interventions: Device: Coronary Sinus Reducer

INTERVENTIONS:
Device: Coronary Sinus Reducer — Implantation of Coronary Sinus Reducer

SUMMARY:
The increasing number of coronary revascularization procedures, coupled with improvements in drug therapy, has significantly extended the lifespan of patients with coronary artery disease (CAD). However, there remains a significant number of CAD patients who experience disability due to chronic refractory angina pectoris. These patients typically have severe diffuse CAD and are not candidates for further revascularization involving surgical coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI).

The installation of a coronary sinus reducer (CSR) represents a new option for percutaneous treatment of patients with refractory angina pectoris who are not suitable for surgical or percutaneous revascularization. The CSR device is designed as an hourglass-shaped stent that is positioned transcatheterally in the distal part of the coronary sinus. This increases intramyocardial venous pressure, which is believed to lead to a more favorable perfusion ratio between the ischemic subendocardial and non-ischemic subepicardial myocardium. Previous research has demonstrated that the implantation of CSR is a safe and relatively straightforward procedure. However, broader implementation and better patient selection are still limited by the fact that the exact mechanism of action remains controversial. It has not been determined why some patients have better outcomes compared to others with seemingly similar coronary artery disease. It is known that patients with atherosclerotic changes in the epicardial coronary arteries also have a certain degree of coronary microcirculation disease (the coronary vascular bed encompassing vessels with a diameter < 200 μm), which cannot be assessed through standard coronary angiography. This study aims to assess changes in coronary microcirculation after the implantation of CSR by measuring coronary flow reserve (CFR) and index of microcirculatory resistance (IMR) before and 6 months after the procedure. Furthermore, our goal is to associate these changes with clinical symptoms and myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease and refractory angina pectoris who are ineligible for coronary revascularization
* Signed informed consent

Exclusion Criteria:

* Severely reduced systolic ejection fraction of the left ventricle (EF < 35 %)
* Severe renal impairment (eGFR < 30ml/min/1.73m2)
* Severe chronic obstructive pulmonary disease (GOLD D)
* Contraindication for application of papaverine or regadenoson

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Impact of Coronary Sinus Reducer on Coronary Microcirculation | 2 and half years
  Assessment of Coronary Flow Reserve and Index of Microcirculatory Resistance before and after Coronary Sinus Reducer implantation

SECONDARY OUTCOMES:
Myocardial Ischemia assessment | 2 and half years
  Evaluation of the ischemic zone before and 6 months after the procedure using Perfusion Stress Cardiac Magnetic Resonance
Angina assessment | 2 and half years
  Comparison of the severity of angina pectoris before and 6 months after the procedure using the Canadian Cardiovascular Society angina scale (CCS) and the Seattle Angina Questionnaire-7 (SAQ-7).
Functional capacity assessment | 2 and half years
  Assessment of functional capacity before and 6 months after the procedure through 6 Minute Walk Test

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia